CLINICAL TRIAL: NCT06307236
Title: Dysmenorrhea of Emotional Freedom Techniques (EFT) and Its Effect on Perceived
Brief Title: Dysmenorrhea of Emotional Freedom Techniques (EFT) and Its Effect on Perceived Stress Level
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Elif TUGCE CITIL, assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-41997688-050.99-105442
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea Primary; Stress; Emotional Freedom

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant
Masking Description: Single Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Group to be applied EFT
  Interventions: Behavioral: Emotional Freedom Techniques
- Control (No Intervention): No application will be made

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques — Emotional Freedom Technique (EFT), which is included in the energy psychotherapy similar to the cognitive behavioral therapy method, is an easily applicable method that is used to relieve mental problems such as anxiety and stress and has positive results, which has just started to be used in the world and in our country. EFT can be applied safely to all ages and groups.
  Arms: Experimental

SUMMARY:
The aim of the study is to determine the effect of EFT application on the level of dysmenorrhea and stress perception in women with dysmenorrhea. For this purpose, EFT will be applied to women with dysmenorrhea with high stress perception assigned to the experimental and control groups, and their stress perceptions and dysmenorrhea levels will be re-evaluated after the application. Perceived Stress Scale (PSS) and Visual Analog Scale (VAS) will be used in the research.

DETAILED DESCRIPTION:
Application of the experimental group The women in the experimental group will be informed about the function, click points and application of EFT through a written material. The EFT application will be explained practically by a certified researcher and the application steps will be followed. Women who underwent EFT will be contacted again within a week or two and asked how they feel and feedback will be received about whether the problem or problems during the first meeting still bother them. By asking women to show how they feel on the SUE scale, the EFT application will be repeated until the woman expresses positive emotions on the SUE scale. The number of EFT applications will be decided according to the woman's condition. After the EFT application is completed, the woman will be re-evaluated with VAS and PSS in the 1st and 2nd months. It will be recorded and reported as perceived stress when assessing The EFT practitioner researcher's certification is S.E.M. It is a certificate with a total scope of 50 hours, including face-to-face training, issued by the Academy considering International Education standards and criteria. The training was given by a trainer with a trainer certificate on EFT. The researcher, who has a nationally and internationally valid certificate, has prepared a guideline in parallel with the training he has received, received expert opinions on the guideline and will carry out its pilot application.

Application of the control group A meeting will be held with the women in the control group at the beginning of the research and information will be given about the study. The researcher will open a WhatsApp group for the women in the control group and follow them to eliminate their lack of information. Throughout the research, women in the control group will continue their routine coping habits regarding dysmenorrhea and perceived stress levels, and this group, like the experimental group, will be re-evaluated with VAS and PSS in the 1st and 2nd months of the research.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-49 years old and single,
* Must be literate and willing to participate in the study,
* There should be no wounds, scars or infections in the area where EFT will be applied.
* The perceived stress level must be high and they must be experiencing dysmenorrhea

Exclusion Criteria:

* There should be no change in menstrual cycle in the last six months,
* There must be no communication problems or illnesses that may prevent work.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since dysmenorrhea is seen only in women, our study will be conducted with women.
Enrollment: 56 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
EFT application | 12 weeks
  Perceived stress scale, VAS
Control | 12 weeks
  Perceived stress scale, VAS

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe ÇİTİL, Principal Investigator — Kütahya Health Science University
Locations (1):
- Kütahya Health Science University, Kütahya, Turkey (Türkiye)